CLINICAL TRIAL: NCT03342703
Title: Correlation of Ultrasound Based Measurements of Liver Stiffness and Steatosis With MRI
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Aya Kamaya, Associate Professor of Medicine, Stanford University
Other Study IDs: 38649
Record Dates: First submitted 2017-10-12; First posted 2017-11-17 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Liver Steatoses; Liver Cirrhosis
MeSH Terms: conditions — Fatty Liver; Liver Cirrhosis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Patients with Liver Fibrosis Measurement: Group1: Patients will undergo an Ultrasound to correlate fibrosis measurements obtained using standard-of-care MRI.
  Interventions: Diagnostic Test: Ultrasound
- Patients with Liver Steatosis Measurement: Group 2: Patients will undergo an Ultrasound to correlate steatosis measurements obtained using standard-of-care MRI.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Patients will undergo a standard liver US protocol for approximately 15 minutes.
  Other Names: US elastography; US fat quantification

SUMMARY:
The investigators will assess the ability of ultrasound (US) to measure liver stiffness (cirrhosis) and liver fat content (steatosis).

DETAILED DESCRIPTION:
Non-invasive monitoring of liver fibrosis using magnetic resonance imaging (MRI) can help determine which patients will most benefit from interventional therapies to help reverse the condition. Similarly, quantitative assessment of liver fat content using MRI can assist physicians in identifying patients at risk for hepatic steatohepatitis.

Due to the widespread dissemination of US machines and their relative lower cost compared to other imaging modalities, e.g. MRI, the ability of US to assess these parameters widens diagnostic availability.

Patients who have undergone an MRI exam to assess liver stiffness (cirrhosis) and/or liver fat content (steatosis) will be asked to undergo an US exam to assess the same parameters. The cirrhosis and steatosis measurements obtained from both exams will be compared. If US-based measurements of liver stiffness and/or liver fat content are shown to be reproducible and accurate when compared to MRI values (will be used as the gold standard), US may become the first-line diagnostic test for these liver conditions.

ELIGIBILITY:
Inclusion Criteria:

1. participants who have a clinical indication for a standard of care MRI exam that included assessment of the liver
2. participant is at least 18 years of age

Exclusion Criteria:

1. Participants unable to take part in the decision making process on whether to consent to the trial
2. Patients with previous chemoembolization or other focal liver therapies to the liver (* NOTE: for liver transplant patients, this criterion is only applicable to the transplanted liver)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have or are scheduled to undergo a routine clinical MRI at Stanford that included assessment of liver stiffness or liver fat content will be identified using the radiology schedule.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Discriminatory value (AUC) of US in assessing liver stiffness | an estimated time of 30 minutes
  Discriminatory value (the ability of the test to diagnose disease from healthy) will be calculated using nonparametric receiver operating characteristic (ROC) curve analysis. Sensitivity (i.e. true positive rate: the ability of a test to correctly identify patients with the disease being investigated) is plotted on the y axis and 1-specificity (i.e. false positive rate: the test incorrectly identifies patients who do not have the disease being investigated as having the disease) will be plotted on the x-axis. Cutoff points of US liver stiffness values will be chosen to create the graph of sensitivity versus 1-Specificity, i.e. the ROC curve, and the area under the curve (AUC) is used to determine how well US discriminates patients with liver stiffness from patients without liver stiffness.
  The closer the AUC gets to 1, the more discriminatory the test. An AUC=0.5 is a test that is right 50% of the time, and is no better than flipping a coin.
Discriminatory value (AUC) of US in assessing liver fat content | an estimated average of 30 minutes
  Discriminatory value (the ability of the test to diagnose disease from healthy) will be calculated using nonparametric receiver operating characteristic (ROC) curve analysis. Sensitivity (i.e. true positive rate: the ability of a test to correctly identify patients with the disease being investigated) is plotted on the y axis and 1-specificity (i.e. false positive rate: the test incorrectly identifies patients who do not have the disease being investigated as having the disease) will be plotted on the x-axis. Cutoff points of US liver fat content values will be chosen to create the graph of sensitivity versus 1-specificity, i.e. the ROC curve, and the area under the curve (AUC) is used to determine how well US discriminates patients with liver fat content from patients without liver fat content.
  The closer the AUC gets to 1, the more discriminatory the test. An AUC=0.5 is a test that is right 50% of the time, and is no better than flipping a coin.

SECONDARY OUTCOMES:
US Elastography Stiffness | an estimated average of 30 minutes
  MRI tissue stiffness is reported in shear modulus (S), while US uses Young's modulus (Y). Since Y = 2*(1+m)*S, where m is the Poisson's ratio for the material, and since that ratio is between 0.49 and 0.50 for tissue, the US measurements should be three times that of the MRI ones. In particular, treating the MRI measurements as the reference, theory predicts a linear relationship:
  Y = 0 + 3*S
  which can be tested with a linear regression model. The most straightforward means is by calculating the expected Young's modulus values for US from the MR measurements, and regressing them on the observed US measurements.
  Both US and MRI values are given below.

CONTACTS AND LOCATIONS:
Overall Officials: Aya Kamaya, MD, Principal Investigator — Stanford University; Andreas Loening, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University Hospital, Stanford, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No